CLINICAL TRIAL: NCT03229265
Title: Pharmacokinetic Study of Tacrolimus and Mycophenolate Mofetil in Kidney Transplant Recipients With Hyperkalemia Receiving Patiromer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1606017355
Record Dates: First submitted 2017-06-12; First posted 2017-07-25 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Hyperkalemia; Kidney Transplant
MeSH Terms: conditions — Hyperkalemia | interventions — patiromer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patiromer (Experimental)
  Interventions: Drug: Patiromer

INTERVENTIONS:
Drug: Patiromer — Patiromer (8.4 grams) will be taken daily at 3 hours after oral tacrolimus and MMF dosing by subjects commencing 3 days (± 1 day) prior to visit 1.

SUMMARY:
Hyperkalemia (high potassium in blood) is a common condition found in kidney transplant patients. Risk factors include poor kidney function and exposure to various drugs. Regardless of the causes, current treatment options are limited. Previously, the only available potassium binder for lowering potassium in the blood is sodium polystyrene sulfonate, which has unknown drug interaction profile with transplant medications. Patiromer is a newly approved potassium binder indicated for the treatment of hyperkalemia. Kidney transplant patients with hyperkalemia may benefit from patiromer. However, the interaction of patiromer and transplant medications has not been studied. The goal of this study is to look into the drug interactions between patiromer and transplant medications.

DETAILED DESCRIPTION:
This is an open-label single center pharmacokinetic study of kidney transplant recipients with hyperkalemia receiving tacrolimus and MMF-based immunosuppression.

Subjects will be screened for inclusion and exclusion criteria during the screening visit. There will be 2 study visits (visit 0 and visit 1) for each subject after successful screening. Visit 0 occurs within 14 days (± 3 days) after screening. Visit 1 occurs at 7 days (± 3 days) after visit 0. There will be 3 clinical visits (standard of care) after visit 1. A total of 6 visits are anticipated for this study.

Standard diet for lunch and dinner will be provided to subjects during visit 0 and visit 1. Meals provided will be monitored in relationship to C0 and C12.

During screening visit, blood tests for baseline BMP, aldosterone, magnesium, tacrolimus, DSA, and MMF will be obtained. If applicable, concomitant fludrocortiosone will be stopped prior to screening.

During visit 0, tacrolimus levels will be drawn immediately before (0 hr) and at 8 intervals after dosing (1,2,3,4,5,6,9,12 hrs). MMF levels will be drawn immediately before (0 hr) and at 9 intervals after dosing (1,2,3,4,5,6,7,9,12 hrs). Basic metabolic profile and serum magnesium levels will be drawn immediately before tacrolimus dosing. Oral MMF and tacrolimus will be dosed at 8am ± 1hr.

Enrollment is defined as the first day when subject receives patiromer treatment. Patiromer (8.4 grams) will be taken daily at 3 hours after oral tacrolimus and MMF dosing by subjects commencing 3 days (± 1 day) prior to visit 1. No tacrolimus or MMF dosing changes are allowed between visit 0 and 1. The addition of new concomitant drugs causing interactions with tacrolimus and MMF are prohibited between visit 0 and 1.

During visit 1, subjects will follow the same protocol of blood draws as visit 0. Tacrolimus levels will be drawn immediately before (0 hr) and at 8 intervals after tacrolimus dosing (1,2,3,4,5,6,9,12 hrs). MMF levels will be drawn immediately before (0 hr) and at 9 intervals after MMF dosing (1,2,3,4,5,6,7,9,12 hrs). Basic metabolic profile and serum magnesium levels will be drawn immediately before tacrolimus dosing. Patiromer at 8.4 grams will be given 3 hrs after tacrolimus and MMF dosing. Oral MMF and tacrolimus will be dosed at 8am ± 1hr.

All subjects will followup for clinical visits (2-4) with the PI or their transplant nephrologists after visit 1 according to schedule (see appendix for study visit events). Subjects will complete study by 30 days (± 7 days) after visit 0. Adjustment of patiromer dosing is at the discretion of PIs after visit 2. After completion of study visits, subjects will continue to follow with transplant clinic monthly for 2 months or sooner if clinically indicated per the discretion of the treating transplant nephrologist. After 2 months, clinic visits will be conducted per routine clinic schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older.
2. Patient is capable of understanding the purposes and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study.
3. Kidney transplant recipient.
4. Must be receiving MMF for maintenance immunosuppression
5. Must be receiving tacrolimus for maintenance immunosuppression
6. Subjects must have hyperkalemia (serum potassium ≥ 5.0 mEq/L and ≤ 6.0 mEq/L).
7. Prior to enrollment, subjects must be taking a steady dose of tacrolimus for 3 days.

Exclusion Criteria:

1. Use of Kayexalate 1 day prior to screening visit.
2. Serum potassium level of greater than 6.0 mEq/L at screening.
3. Serum magnesium level of less than 1.0mg/dL at screening.
4. Acute rejection episode within 30 days prior to enrollment.
5. Anemia with hemoglobin level of ≤ 9.0 g/dL prior to screening.
6. Patient has hypersensitivity to patiromer.
7. Receiving maintenance corticosteroid for immunosuppression
8. Serious medical (including history of cardiac arrhythmias) or psychiatric illness likely to interfere with participation in this clinical study.
9. Patients with known donor-specific antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
AUC | Within 30 days
  Investigate the pharmacokinetics of tacrolimus and mycophenolate mofetil in kidney transplant recipients receiving patiromer. Investigators will obtain serum levels of tacrolimus and mycophenolate mofetil before and after the administration of the study drug patiromer. Investigators will measure the areas under the curve of tacrolimus and mycophenolate mofetil before and after exposure to patiromer.

SECONDARY OUTCOMES:
Serum potassium levels | Within 30 days
  To assess the effect of patiromer in reducing hyperkalemia. Investigators will measure the serum potassium levels after the administration of the study drug patiromer.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Lee, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided